CLINICAL TRIAL: NCT05990933
Title: Role of Adrenaline in the Inflammatory Response in People with Diabetes Mellitus Type 1, and Healthy Individuals
Brief Title: Role of Adrenaline in in the Inflammatory Response in Diabetes
Acronym: RAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cees Tack (Other)
Responsible Party: Sponsor-Investigator, Cees Tack, Prof. Dr., Radboud University Medical Center
Organization: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 114664
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Response; Diabetes Type1; Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — Epinephrine

STUDY DESIGN:
Intervention Model Description: All participants will receive intravenous infusion of adrenaline at a rate of 0.04ug/kg/min for 1 hour. We will draw blood at baseline, 30 minutes, 60 minutes, 180 minutes, 24 hours 72 and a week after start of infusion. These samples will be used for phenotyping of the innate immune system and measuring inflammatory and atherogenic parameters. Throughout the infusion vital parameters will be monitored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- People with type 1 diabetes (Experimental): The participants with type 1 diabetes will receive an intravenous infusion of adrenaline at a rate of 0.04ug/kg/min for 1 hour.
  Interventions: Drug: Adrenaline
- Healthy individuals (Active Comparator): The participants without type 1 diabetes will receive an intravenous infusion of adrenaline at a rate of 0.04ug/kg/min for 1 hour.
  Interventions: Drug: Adrenaline

INTERVENTIONS:
Drug: Adrenaline — Adrenaline infusion at a rate of 0.04ug/kg/min for 1 hour administered intravenously.
  Other Names: Adrenaline infusion

SUMMARY:
The primary aim of the present study is to study the effect of adrenaline administration on inflammatory parameters (e.g. leukocyte phenotype, cytokines, inflammatory proteins). Secondary objectives consist of the effect of adrenaline on atherogenic parameters.

* All participants will receive intravenous infusion of adrenaline for an hour
* We will draw blood at 7 time points, not including screening
* Participants will be asked to return for a total of 4 times

Researchers will compare 2 groups, healthy individuals versus people with diabetes type 1 to see if the inflammatory reaction to adrenaline differs between these two groups.

DETAILED DESCRIPTION:
Objective: The aim of the present study is to study the effect of increased adrenaline levels on the inflammatory response (e.g. leukocyte phenotype, cytokines, inflammatory proteins) by administering exogenous adrenaline in participants with type 1 diabetes and healthy participants.

Potentially eligible adult ( 16 - 75 years) participants will be recruited from the diabetes clinic at the department of internal medicine from the Radboud University Medical Center. Healthy participants will be recruited through social media and other advertisements. We will recruit a total of 30 individuals, i.e. 15 healthy participants and 15 people with type 1 diabetes. Participants with type 1 diabetes will be equipped with a blinded continuous glucose monitoring device (CGM) during the test, which will measure interstitial glucose levels for a total of 10 days.

Intervention: All participants will receive intravenous infusion of adrenaline at a rate of 0.04ug/kg/min for 1 hour. We will draw blood at baseline, 30 minutes, 60 minutes, 180 minutes, 24 hours 72 hours and a week after start of infusion. The blood samples will be used for phenotyping of the innate immune system and measuring inflammatory and atherogenic parameters. Throughout the infusion, vital parameters will be monitored.

ELIGIBILITY:
Overall inclusion criteria:

* Ability to provide written informed consent
* Body-Mass Index: 19-30kg/m2
* Age ≥16 years, ≤ 75 years
* Blood pressure: <140/90 mmHg
* Non-smoking
* Electrocardiogram not showing any serious arrythmia's (PVC's and PAC's accepted)

Diabetes group specific criteria:

* Insulin treatment according to basal-bolus insulin regimen (injections or insulin pump)
* Duration of diabetes > 1 year
* HbA1c < 100 mmol/mol,

Exclusion Criteria:

* Any event of cardiovascular disease in the past 5 years (e.g. myocardial infarction, stroke, heart failure, symptomatic peripheral arterial disease)
* Pregnancy or breastfeeding or unwillingness to undertake measures for birth control
* Epilepsy
* Current treatment with Alpha or beta blockers ( doxazosin, propranolol)
* History of panic disorders
* History of Arrhythmias
* Use of immune-modifying drugs or antibiotics
* Use of tricyclic antidepressants or MAO inhibitors
* Use of statins (e.g. stop statins >2 weeks before performing blood sampling.
* Any infection with systemic symptoms in past 2 weeks
* Previous vaccination in the past 2 weeks
* Proliferative retinopathy
* Nephropathy with an estimated glomerular filtration rate (by MDRD) ˂60ml/min/1.73m2

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Monocyte count | Change from baseline compared to after 1 hour
  The amount of monocytes following 60 minutes of adrenaline infusion compared to baseline to asses the adrenaline effect on the inflammatory response.

SECONDARY OUTCOMES:
Leukocyte count | Change from baseline at day 30, 60 and 180 minutes 1, day 3 and day 7 after adrenaline infusion
  Measurement of the amount of leukocytes
Leukocyte phenotype | Change from baseline at day 30, 60 and 180 minutes 1, day 3 and day 7 after adrenaline infusion
  Measuring several phenotypes by using a pre-defined panel of interest with flow-cytometry ( e.g. NK-cells, granulocytes)
Pro-inflammatory proteins | Change from baseline at day 30, 60 and 180 minutes 1, day 3 and day 7 after adrenaline infusion
  Pro-inflammatory proteins using Olink Proteomics AB inflammation panel with 92 circulating inflammatory proteins ( e.g. EN-rage, FIT3L)
Inflammation plasma parameters | Change from baseline at 30, 60 and 180 minutes day 1, day 3 and day 7 after adrenaline infusion
  Inflammatory plasma protein using ELISA, ( e.g high sensitive-crp)
Atherogenic parameters | Change from baseline at 30, 60 and 180 minutes day 1, day 3 and day 7 after adrenaline infusion
  Atherogenic parameters using ELISA method including but not limited to, VCAM-1, ICAM-1, E-Selectin, P-selectin, PAI-1, Plasma Endothelin
Insulin | Change from baseline at, 60 and 180 minutes
  Plasma levels of insulin
Adrenaline | Change from baseline at 30, 60 and 180 minutes
  Plasma levels of adrenaline
Noradrenaline | Change from baseline at 30, 60 and 180 minutes
  Plasma levels of noradrenaline
Glucose variability | 2 weeks
  Glucose variability measured by the blinded continuous glucose monitor including but not limited to, measuring time within range, amount of hypoglycaemic events, amount of hyperglycaemic events.
Ex vivo cytokines | Change from baseline at 30, 60 and 180 minutes, day 1, day 3 and day 7 after adrenaline infusion
  Ex vivo production of pro- and anti-inflammatory cytokines and chemokines after ex vivo stimulation of isolated monocytes, including TNF-α, IL-6, IL-10 and IL-1β.
Distribution of monocyte subset | Change from baseline at 30, 60 and 180 minutes, day 1, day 3 and day 7 after adrenaline infusion
  Distribution of pro- and anti-inflammatory monocyte subsets using FACS (Fluorescence-activated Cell Sorting)

CONTACTS AND LOCATIONS:
Overall Officials: Cees Tack, MD. PHD., Principal Investigator — Radboud University Medical Center (Radboudumc)
Locations (1):
- Radboud UMC, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
WE will share the study protocol using a data respository accesible through the research team on demand. Starting around 6 months after publication.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: The coordinating researcher will review acces requests. Seeing as the data are all anonimised acces will be granted for additional research in the field of inflammation or diabetes.

REFERENCES:
- [Derived] Mustafajev IF, Hendriksz MS, Stienstra R, Tack CJ, de Galan BE, Meijer RI. Adrenaline is a prominent driver of inflammatory responses following hypoglycaemia. Diabetologia. 2026 Jan 29. doi: 10.1007/s00125-026-06667-9. Online ahead of print. PMID 41611977